CLINICAL TRIAL: NCT00047957
Title: The Effect of Peripheral Homotopic and Heterotopic Stimulation on Cortical Excitability
Brief Title: Brain Inhibition of Muscle Movement in Normal Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030008; 03-N-0008
Record Dates: First submitted 2002-10-22; First posted 2002-10-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: Dystonic Disorders
Keywords: Transcranial; Magnetic; Stimulation; Motor; Cortex; Motor Cortex; Afferent Stimulation; Transcranial Magnetic Stimulation; Healthy Volunteer; HV
MeSH Terms: conditions — Dystonic Disorders

SUMMARY:
This study will use transcranial magnetic stimulation, or TMS (described below), to examine how the brain controls muscle movement to prevent unwanted movements in surrounding muscles. For example, when a person moves a finger, a part of the brain called the cortex prevents unwanted movements in other fingers by a process called cortical inhibition. In people with the muscle disorder dystonia, cortical inhibition does not work properly and patients suffer from uncontrolled and sometimes painful movements. A better understanding of how this process works in normal people may shed light on what goes wrong in dystonia and how the condition can be treated.

Healthy normal volunteers 19 years of age and older may be eligible for this study. Candidates will be screened with a medical history and physical and neurological examinations. People with a current medical or surgical condition or neurological or psychiatric illness may not participate, nor may individuals who are taking medication that may influence nervous system function.

Participants will undergo TMS to record the electrical activity of muscles in the hand and arm that are activated by magnetic stimulation. For the procedure, subjects are seated in a chair with their hands placed on a pillow in their laps. A wire coil in placed on their scalps. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. Subjects will be asked to move their second finger in response to a loud beep or visual cue. In some trials, a brief, mild electrical shock will also be applied to the end of either the second or fifth finger. The shock is not painful.

TMS may cause muscle, hand or arm twitching if the coil is near the part of the brain that controls movement, or it may induce twitches or temporary tingling in the forearm, head, or face muscles. The twitching may cause mild discomfort, but the procedure is rarely considered painful.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of homotopic and heterotopic sensory afferent input on surround inhibition in the motor cortex. Surround inhibition is a cortical phenomenon, the function of which may be to suppress unwanted movements in surrounding muscles during voluntary actions. In support of this, a recent study showed that motor output to the little finger was reduced during self-paced, voluntary movements of the index finger, despite an increase in spinal excitability. Work has also shown that in relaxed muscle, homotopic and heterotopic peripheral stimulation results in time dependent modulation of motor cortical excitability. However, no studies have examined the relationship between volitional movement and afferent sensory input on cortical surround inhibition. Therefore, the aim of this study is to examine the changes in surround inhibition when electrical stimulation is applied to either the finger being actively moved (homotopic stimulation) or a separate finger not involved in the movement (heterotopic stimulation) at different time periods prior to the initiation of movements to assess the affect of these stimuli on surround inhibition and excitation in the motor cortex.

ELIGIBILITY:
INCLUSION CRITERIA:

Twenty healthy volunteers older than age 18 will be recruited for the study. Their gender, age, or ethnic origin will not provide bias for inclusion to the study. All subjects will sign an informed consent prior to participation in the trial.

EXCLUSION CRITERIA:

Exclusion criteria for the trial will include any current medical or surgical condition or neurological or psychiatric illnesses. Furthermore, any individual who is on medication with potential influence on nervous system function, who has a pacemaker, an implanted medical pump, a metal plate or metal object in the skull or eye (for example, after brain surgery), or who has a history of seizure disorder will be excluded from the trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2002-10; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Abbruzzese G, Marchese R, Buccolieri A, Gasparetto B, Trompetto C. Abnormalities of sensorimotor integration in focal dystonia: a transcranial magnetic stimulation study. Brain. 2001 Mar;124(Pt 3):537-45. doi: 10.1093/brain/124.3.537. PMID 11222454
- [Background] Classen J, Steinfelder B, Liepert J, Stefan K, Celnik P, Cohen LG, Hess A, Kunesch E, Chen R, Benecke R, Hallett M. Cutaneomotor integration in humans is somatotopically organized at various levels of the nervous system and is task dependent. Exp Brain Res. 2000 Jan;130(1):48-59. doi: 10.1007/s002210050005. PMID 10638440
- [Background] Hallett M. Transcranial magnetic stimulation and the human brain. Nature. 2000 Jul 13;406(6792):147-50. doi: 10.1038/35018000. PMID 10910346